CLINICAL TRIAL: NCT00256581
Title: Imaging Studies With GE C-Hawk Gamma Camera Compared to Routine Clinical Exam
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Other Study IDs: 2005-0273
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease; Chest Pain
Keywords: myocardial perfusion; Imaging
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Additional rest and stress image sets on new camera

SUMMARY:
Comparison study of myocardial perfusion SPECT imaging with current clinical use camera and new camera.

DETAILED DESCRIPTION:
Comparison study of myocardial perfusion SPECT imaging with current clinical use camera and new camera.

ELIGIBILITY:
Inclusion Criteria:

* Referral for cardiac stress testing with SPECT myocardial perfusion imaging

Exclusion Criteria:

* refusal to provide written informed consent or lack capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing SPECT Myocardial perfusion imaging
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hellman, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health, Madison, Wisconsin, United States